CLINICAL TRIAL: NCT03558919
Title: Efficacy and Safety of Mirabegron Compared With Solifenacin in Treatment of Overactive Bladder
Brief Title: Efficacy and Safety of the Mirabegron Compared With Solifenacin in Treatment of Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. A S M Kutub Uddin Awal, Final year Resident, Department of urology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mirabegron
Record Dates: First submitted 2018-04-18; First posted 2018-06-15 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Intervention Model Description: Randomized Controled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Mirabegron (Experimental): Mirabegron 25mg will give daily at night for 12 weeks
  Interventions: Drug: Mirabegron 25mg
- Solifenacin (Active Comparator): Solifenacin Succinate 5mg will give daily at night for 12 weeks
  Interventions: Drug: Solifenacin Succinate 5 MG

INTERVENTIONS:
Drug: Mirabegron 25mg
  Arms: Mirabegron
Drug: Solifenacin Succinate 5 MG
  Arms: Solifenacin

SUMMARY:
Overactive bladder (OAB) is a chronic symptom complex that can substantially impair quality of life. Pharmacological management using antimuscarinics agent remain the mainstay of therapy and effectively reduce OAB symptoms. However, despite the proven efficacy of such agents, their tolerability may be limited by adverse events, mostly dry mouth. In fact these adverse events often lead to poor compliance and discontinuation of therapy.The β3-adrenoceptor agonist, mirabegron, which acts via a different mechanism of action to antimuscarinics, could potentially improve the efficacy/ tolerability balance over current standard of care in the management of OAB.β3-adrenoceptor agonists relax detrusor smooth muscle during the bladder storage phase and increase bladder capacity without negatively affecting voiding parameters. Different study has report efficacy and safety of mirabegron but not done in our country.

Investigators will evaluate the efficacy and safety of mirabegron comparison with solifenacin succinate in the treatment of overactive bladder.This is a hospital based prospective randomized controlled clinical trial will be conducted from July 2016 to November 2017 in the department of urology, Bangabandhu Sheikh Mujib Medical University (BSMMU). Among the patient with overactive bladder who will visit to Urology outpatient department (OPD) of BSSMU, 56 patient who will fulfil the inclusion criteria will be selected. Selected patients will be evaluated by history, physical examinations and investigation like routine urine analysis & culture, serum creatinine, random blood sugar, X-ray kidney, ureter & bladder (KUB) region,ultrasonogram (USG) of KUB region with maximum cystometric capacity (MCC) & post-viodal residue (PVR). After taking informed consent, selected 82 patient will be randomly divided in to experimental group and control group, each containing 41 patients. All patients will be entered into one week run-in period, when they will instructed to stop any drug including any anti-cholinergics, if they are getting it before. Patient will be supplied with a Bengali version micturition diary from and instructed to complete a 3 day voiding diary. Average of three day will be calculated for 24 hours.Overactive symptom score will be calculated by interviewing the patient for urinary symptom for last 7 days. Experimental group will receive Mirabegron 25mg and control group will receive solifenacin succinate 5 mg all are at night for 12 weeks. Patients in both group will be regularly followed up 12 weeks at 4 weeks interval.Patient will be supplied with a Bengali version micturition diary from and instructed to complete a 3 day voiding diary in each follow up schedule visit at the end of 4, 8 and 12 weeks. Overactive symptom score will be calculated by interviewing the patient for urinary symptom for last 7 days in each visit.Patient will be evaluated for any adverse effects during the medication. Data will be collected, complied, computed and appropriate statistical analysis will be done as per objectives

DETAILED DESCRIPTION:
Introduction:

Overactive bladder syndrome (OAB) is defined by the International Continence Society as urinary urgency, with or without urgency incontinence, usually with increased daytime frequency and nocturia in the absence of proven infection or any other pathology.

Epidemiological data suggest that OAB syndrome is present in about 10.7% of all adult men and women, although prevalence rates increase with aging in both sexes. The prevalence of OAB worldwide is estimated as being greater in women versus men (11.6% vs 9.7%, respectively) It is a chronic symptom complex that can substantially impair quality of life. The prevalence of lower urinary tract symptom (LUTS), OAB and urgency urinary incontinence is substantial, affecting both women and men, and resulting in considerable morbidity, personal cost and health economic burden.

Initial management uses conservative measures, such as fluid advice and bladder training.

Antimuscarinic drugs (eg. Solifenacin succinate) are still the mainstay of oral pharmacological treatment for OAB, relaxing the detrusor muscle and reducing sensory symptoms during the storage phase of the micturition cycle by inhibiting muscarinic receptor subtypes, M2 and M3. Both subtypes are expressed in multiple tissues, increasing the risk of bothersome, anticholinergic adverse events (AEs) such as dry mouth, which along with lack of efficacy, is the most frequently cited reason for discontinuation of antimuscarinic treatment.

Recent advances in the understanding of OAB have identified three β-adrenoceptor sub-types β1, β2 and β3, in the detrusor muscle and urothelium .The β3-adrenoceptor is the predominant β-receptor subtype in the human urinary bladder.

β3-adrenoceptor agonists relax detrusor smooth muscle during the bladder storage phase and increase bladder capacity without negatively affecting voiding parameters, including maximum urinary flow rate (Qmax), detrusor pressure at Qmax (PdetQmax), and residual volume.

The β3-adrenoceptor agonist, mirabegron, which acts via a different mechanism of action to antimuscarinics, could potentially improve the efficacy/ tolerability balance over current standard of care in the management of OAB. In four 12-week phase III studies mirabegron consistently demonstrated superiority over placebo with respect to reductions in incontinence episodes and micturition frequency.

The main adverse effects of mirabegron is hypertension, nasopharyngitis, headache and urinary tract infection. Dry mouth and constipation are similar as placebo but lower than the solifenacin succinate.

There were several studies observe mirabegron is effective as well as well tolerable in OAB. There was a single comparative study between mirabegron & solifenacin shows non inferiority of mirabegron than solifenacin. But all the study done by industrial sponsored. In Bangladesh, no such study was performed previously. So it is time demanding to conduct a comparative study between the safety and efficacy of mirabegron & solifenacin in patient with overactive bladder in this country.

This new drug β3 adrenoceptor agonist mirabegron is available as 25mg once daily formulation in the treatment of OAB in Bangladesh.

This study has been designed to see the efficacy and safety of mirabegron comparison with solifenacin succinate in the treatment of overactive bladder without industrial support.

Hypothesis Null hypothesis (H0): There is no difference in efficacy and safety of mirabegron and solifenacin succinate for treatment of overactive bladder.

Alternate hypothesis (HA):The efficacy and safety of mirabegron is superior to solifenacin succinate for treatment of overactive bladder.

Objective General objective To compare the therapeutic efficacy and safety of mirabegron comparison with solifenacin succinate in the treatment of overactive bladder.

Specific objective

* Compare the overactive bladder symptom score (OABSS) between both treatment group.
* To find out the micturition frequency and nocturia of the both treatment group and compare between them.
* To find out the urgency and urge incontinence of the both treatment group and compare between them.
* To compare the adverse effects of mirabegron and solifenacin succinate to treat overactive bladder.

Methodology:

Type of study: Hospital based prospective randomized controlled clinical trial.

Study period: July 2016 to November 2017.

Place of study: Department of Urology, Bangabandhu Sheikh Mujib Medical University(BSMMU), Dhaka, Bangladesh.

Study subject:

Men and women age at least 18 years with persistent overactive bladder (OAB) symptoms for 3 months or more and will be treated as out patients who attended in the out patient department of Urology, BSMMU, Dhaka, will be enrolled in this study.

Sampling technique:

Purposive sampling technique will be applied to collect the sample for this study.

The patent will come with the symptoms of OAB in outpatient department of urology of BSMMU hospital will be selected as per inclusion and exclusion criteria for the present study. After written informed consent, a total 82 will be recruit and divided into two groups by randomization. First participant will selected by lottery method then rest of the participants will be enrolled alternatively dividing into two groups.

Methods This randomized clinical will be conduct in the department of urology, BSMMU, Dhaka after receiving approval from Institutional Review Board (IRB). The study population will select on the basis of selection criteria from the patient attended in the out patient department of Urology, BSMMU, Dhaka.

Evaluation of patients before drug therapy:

Study commence with the initial visit during which a complete medical history was taken along with a physical examination with special attention to uro-genital and nervous system. Digital rectal examination (DRE) will be done to exclude any suspected pelvic pathology causing bladder outlet obstruction (BOO) and neuropathic bladder by assessing perianal sensation and anal tone, bulbocavernous reflex and other relevant neurological examination.

Laboratory screening for Hb% and clinical chemistry (blood sugar, serum creatinine) and urine routine examination and culture and sensitivity will be done to exclude urinary tract infection (UTI). Ultrasonography of the KUB region with MCC and PVR will be done to exclude any obstructive uropathy. Plain x-ray KUB will be done to exclude urinary stone disease and any lesion in vertebral column.

After complete of baseline clinical evaluation and investigation, those meting the inclusion criteria will be selected for the present study.

A written informed consent will be taken from all the study subject without exploiting any of their weakness. For the study a well-informed, voluntary, signed written consent will be taken in an understandable local language from the patient after convincing them that their privacy and confidentiality will be safeguard.

A data sheet will be complete for each patient included particulars of the patient, relevant history, examination finding and relevant baseline investigation.

All patients will be entered into one week run-in period, when they will instructed to stop any drug including any anti-cholinergics, if they are getting it before. Patient will be supplied with a Bengali version micturition diary from and instructed to complete a 3 day voiding diary. Average of three day will be calculated for 24 hours.

Overactive symptom score will be calculated by interviewing the patient for urinary symptom for last 7 days.

The data sheet will be filled up after taking a brief interview of 15-20 minutes from the patient.

Follow-up:

Patient in both group will be regularly followed up 12 weeks at 4 weeks interval.

Patient will be supplied with a Bengali version micturition diary from and instructed to complete a 3 day voiding diary in each follow up schedule visit at the end of 4, 8 and 12 weeks of treatment to record the number of micturition, urgency, urge incontinence, nocturia, the number of pad used, and voided volume of each micturition / 24 hours over 3 consecutive days. Average of three day will be calculated for 24 hours.

Overactive symptom score will be calculated by interviewing the patient for urinary symptom for last 7 days in each visit.

Patient will be evaluated for any adverse effects during the medication like dry mouth, constipation, blurring vision, hypertension and headache that either intervention can cause also be recorded in the predesigned data collection sheet. Severity of each of the adverse effect will be assess as mild, moderate and severe.

Patient who will discontinue the drug will be excluded from data analysis. All patient will contracted over telephone as schedule visit for follow up after initial treatment.

Technique of voiding diary:

Instruction for completing the 3-days voiding diary Please complete the voiding diary for a total of 3 days. On the day that you start recording events in the voiding diary, print Participant name and date at the top of the diary.

Start a new page for each day you keep the diary. Participant need to keep a diary for 3 full consecutive days.

Measurement of functional improvement after intervention:

It will based on changes in the number of micturitions, urgency, and urge incontinence episodes, nocturia episodes, the number of pad used, the voided volume of each micturition, per 24 hours and OABSS after 4, 8 and 12 weeks of drug intervention. This record will compare with baseline record.

Data Processing Plan:

Data collection instrument:

Data collection sheet Title:Efficacy and safety of mirabegron compared with solifenacin in treatment of overactive bladder Name of the investigator: Dr. A. S. M. Kutub Uddin Awal Place of study: Department of urology, BSMMU, Shahbag Dhaka.

Particulars of the patient:

Serial no……………………………. Date……………. Name………………………………………………………. Age……………… Sex:-Male/Female Telephone no……………...................

Address:- Present ……………………………………………………………… ………………………………………………………………………

Group:

1. Mirabegron
2. Solifenacin Succinate

Presenting complaints:

1. Micturition frequency per 24 hours…………………………………….
2. Episodes of urgency per 24 hours………………………………………
3. Urge incontinence episodes per 24 hours……………………………..
4. Nocturia…………………………………………………………………….
5. Voided volume of each micturition (ml)…………………………………
6. Overactive bladder symptom score (OABSS) …………………………

Associated co-morbidity:

1. No
2. Diabetes mellitus
3. Hypertension
4. Stroke

Physical examination:

1. Pulse ………b/min,
2. BP…(mm Hg)

1. <139 and/or <90 2. 140-159 and/or 90-99 3. 160-179 and/or 100-109 4. ≥180 and/or ≥110

Investigations:

Hemoglobin ……………………gm/dl Random Blood Sugar ………….. mmol/l. Serum Creatinine …………mg/dl Urine R/M/E Pus cells: 1= 0-4/HPF 2=≥ 5 HPF RBC: 1= 0-3/HPF 2=>3/HPF Urine Culture: 1= Positive 2=Negative USG of KUB&P with MCC and PVR: MCC= PVR= Follow up: (from voiding dairy) 4 Weeks 8 Weeks 12 Weeks

1. Micturition frequency per 24 hours
2. Episodes of urgency per 24 hours
3. Urge incontinence episodes per 24 hours
4. Nocturia episodes per 24 hours
5. Voided volume of each micturition (ml)
6. Overactive bladder symptom score (OABSS)

Adverse events:

4 Weeks 8 Weeks 12 Weeks Dry mouth Constipation Blurred vision Headache Hypertension Discontinuation of medication due to adverse events Signature of the investigator

Data Collection:

The demographic information, relevant history, examination findings and investigation reports and outcome of treatment of all the study subjects will be recorded in the data collection sheet.

Patient will be supplied with a Bengali version micturition dairy from and instructed to complete a 3-days voiding dairy prior to medication and each scheduled visit at week 4, 8 and 12 to record the micturition frequency, the presence of urgency and urge incontinence, nocturia episodes, the number of pads used and the voided volume of each micturition. Average of three day will be calculated for 24 hours.

Overactive symptom score will be calculated by interviewing the patient for urinary symptom for last 7 days prior to medication and each scheduled visit.

Any adverse effect during the medication like Dry mouth, Constipation, Blurred vision, Headache and Hypertension that can cause either intervention will be recorded in predesigned data collection sheet.

Patient who will discontinue the drug will be excluded from data analysis. All patient will be contracted telephone as scheduled for follow up after initial treatment.

The data sheet will fill up after taking a brief interview, review of records and documents from the patients.

Data processing and analysis:

Data editing cleaning and reduction will be done by taking care for omission and illegal entry of data. After compilation the data will present in the form of tables and figures as necessary. After data collection all quantitative data will be expressed as mean ± standard deviation and all categorical data will be presented as frequency. Variable will be compared between the groups by Chi- squared test for qualitative variable (frequency, nocturia, urgency) and two sample Z- test for quantitative variable (Overactive symptom score). The statistical software SPSS Statistics version 19 (SPSS ,Chicago Illinois) will be used for statistical analysis of data. Results will be considered significant if p-value <0.05.

Ethical implication:

Ethical clearance for the study will be taken from the Institutional Review Board (I.R.B) of BSMMU prior to the commencement of this study.After the research protocol is approved by the committee, permission for the study will be taken from the Department of Urology, BSMMU. The aims and objectives of the study along with its procedure, risks and benefits of this study will be explained to the study subjects in an easily understandable local language. A written informed consent will be taken from all the study subjects without exploiting any of their weakness. All the study subjects will be assured of adequate treatment of any complications developed in relation to the purpose of the study. All the study subjects will be assured about their confidentiality and freedom to withdraw themselves from the study at any time.

Quality assurance strategy:

During the study period quality assurance strategy will be maintained in every step by meticulous conduct of study and avoidance of any bias. Patient will be select based upon inclusion and exclusion criteria. Before drugs intervention proper counseling will be done with patients regarding the procedure, possible complication and their management. Data collected using questionnaire.

Operational definition:

Overactive bladder syndrome (OAB): Overactive bladder syndrome (OAB) is defined by the International Continence Society as urinary urgency, with or without urgency incontinence, usually with increased daytime frequency and nocturia in the absence of proven infection or any other pathology.

Detrusor over activity (DO): It is an urodynamic observation characterized by involuntary detrusor contraction during the filling phase which may be spontaneous or provoked and is the cause of overactive bladder.

Frequency of micturition: The term is used to describe the need to urinate more often than usual. In this study frequency of micturition will considered 8 or more voids per 24 hours.

Urgency: It is the complaint of a sudden compelling desire to pass urine which is difficult to defer.

Urge incontinence: It is the complaint of involuntary leakage of urine, usually preceded by urgency.

Nocturia: It is the complaint that the individual had to wake at night one or more times to void.

Voided volume of each micturition: It is the volume of urine expelled via urethra in each micturition.

Pad usage: The number of pads are use over 24-hours duration in patient with OAB.

Voiding dairy: It is use for assessing the number of micturitions, present of urgency and urge incontinence, nocturia episodes, pads usage, and voided volume of each micturition. Here, instructed of the patient to complete the 3-days voiding dairy prior to medication and each scheduled visit. (Appendix-) Overactive Bladder Symptom Score (OABSS): This is a single symptom score that employs a self-report questionnaire to quantify OAB symptom. The selected symptom are- day time frequency, nighttime frequency, urgency and urgency incontinence for the questionnaire. Overall score is the simple sum of the four symptom score. (Appendix-)

Informed Consent Form Title:efficacy and safety of mirabegron compared with solifenacin in treatment of overactive bladder

Introduction:

I, Dr. A. S. M. Kutub Uddin Awal, work as student Master of Surgery(MS) (Urology) in the Urology department of Bangabandhu Sheikh Mujib Medical University, Dhaka. Investigators are researching on the treatment of overactive bladder disease that usually impinges on citizens of adult age group. Participants are evocated to provide necessary information about it and participate in our research.

The intention of this 'informed consent form' is to provide participant necessary information that will help you take decision on whether you will participate in this research or not. Participant will not have to take the decision right now. Participant can discuss with anyone before you take the decision.

Aim and methods:

The aim of this 'informed consent form' is to return normal condition of overactive bladder by alone oral medication without any operation.

This research will be conducted by the department of urology, Bangabandhu Sheikh Mujib Medical University. For this research, 82 patients with overactive bladder will be included for the study who will attend in the out patient department of Urology, Bangabandhu Sheikh Mujib Medical University Hospital, Dhaka. There are two types of medication in this study to treat overactive bladder. One of them, you will be taken one tablet in oral once daily. You will have to come back to your physician in every 4 weeks for 3 times, to know the result of research. You will be instructed to complete consecutive 3-days your voiding dairy prior to each follow up scheduled visit. You will be first visited to the investigator at 4 weeks, second time at 8 weeks and last scheduled visit at 12 weeks of treatment period.

If you participate in this study, then we will enroll you in our study and you will be informed everything in details by your physician.

Risk in the research:

In this research participant may have to face a bit risk which is similar to that in case of other medication. The most common harms of the study are dry mouth, constipation, blurred vision, headache, and hypertension. But this risk are very little in favor of your proper treatment. This harm develop in a few patients and usually control without treatment. There is, however, provision for proper treatment of all kinds with appropriate physicians and all necessary facilities within the hospital.

The benefit of participant in the research:

Participant will personally be benefited by your participation in this research. For example, you will receive a more successful treatment option and quickly get free from your symptoms and improvement of quality of life. At the same time, participant will be provided as pioneer to take new treatment option.

Alternative:

The normal treatment of participant will proceed as per the general treatment procedure of the hospital, even if participant do not participate in the research.

Expenditure:

To participant in this research, neither participant will have to carry an additional expenditure nor you will be paid any amount of money.

Confidentiality:

All the information of the research will be kept confidential during the research and afterwards. For the ease of the research you will be given one identification (ID) number. All kind of documents with you ID number will be locked in file cabinet of the office. The personal issue will not be second handed for data analysis, reporting and publishing and will not be disclosed to anyone apart from the examiner of the research. So no one else can be acquainted with any of your information.

Voluntary participation:

The participation of participant in this research is totally voluntary. Participant can deny participating in the research or during the research you can withdraw yourself from the research anytime you want. Your treatment will not be differentiated for that. None of legal right will be breached if you sign this document.

Questionnaire:

Please let us know if participant have any question. We will try to answer your question at our level best. If participant feel like throwing any question in future, then you may contact with researcher Dr. A.S.M. Kutub Uddin awal, department of Urology, Room no 430, Block no-C, Bangabandhu sheikh Mujib Medical University Hospital, Shahbag, Dhaka.

Consent of affirmation:

I am expressing my satisfaction after discussion and with the doctor (the doctor who will do physical examination and the treatment of me) regarding this research. I have understood that my participation in the research is voluntary and I can restrain myself from this research anytime I want without being liable for anything. I have read the above mentioned information / the above mentioned information have read in front of me and I willingly express my affirmation to participate in this research.

Name of the participant:

The Signature of the participant:

Date:

In case of the illiterate participant:

I am testifying that this consent form has read in front of the participant correctly and the participant has the opportunity to ask question. I am confirming that the participant is completely free and consciously agreed to participant in the research.

Name of the witness: The thumb print of the participant:

Signature of the witness:

Date:

.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged ≥18 years
* Patients persistent with OAB symptoms ≥3 months
* The patient able to complete the 3 days voiding diary correctly
* An average of ≥8 micturitions per 24 hours
* An average ≥1 urgency episode per 24 hours
* An average ≥1 nocturia episode per 24 hours

Exclusion Criteria:

* Clinically significant stress or mixed urinary incontinence.
* Abnormal detrusor activity with known neurological diseases.
* Pregnant and lactating women or those who intended to become pregnant during the study.
* Clinically significant bladder outflow obstruction (PVR >100ml), symptomatic urinary tract infection, bladder stones, diabetic neuropathy.
* Significant hepatic, renal or other medical diseases.
* Previous pelvic radiation therapy and malignant disease of the pelvic organs.
* Patients with any condition that contraindicate the use of mirabegron or solifenacin medication (urinary retention, uncontrolled narrow angle glaucoma).
* Patient has severe uncontrolled hypertension, which is defined as a sitting average systolic blood pressure ≥ 180 mm Hg and/ or average diastolic blood pressure ≥ 110 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Overactive symptom score (OABSS) | 12 weeks
  Overactive bladder symptom score Patients are instructed to circle the score that best applies to their urinary condition during the past week; the overall score the sum of the four scores.
  Ques-1 How many times do youtypically urinate fromwaking in the morninguntil sleeping at night? Ques 2 How many times do you typically wake up to urinate from sleeping at night until waking in the morning? Ques 3 How often do you have a sudden desire to urinate, which is difficult to defer? Ques 4. How often do you leak urine because you cannot defer the sudden desire to urinate? Total score Sum of 4 question, Maximum score 15. Reduction OABSS will calculated from baseline

SECONDARY OUTCOMES:
Frequency of micturation | 12 weeks
  Frequency of micturation will be reduced at end of treatment at 12 week calculated from before treatment.
Urgency | 12 weeks
  The percentage of patients with a change from baseline to the final visit in the urgency episodes per 24 hours by 2 or greater.
Urgency incontinence | 12 weeks
  Net change of the mean number of urgency incontinence episodes from baseline to the final visit
Nocturia | 12 weeks
  The net change of mean number of nocturia episodes per 24 hours from baselinev to the final visit
Adverse effects | 12 weeks
  Dry mouth, constipation, blurred vision, hypertension, haedache, nasopharyngitis.
  Number of participant will be developed advers effect during study period will compared between them.
Discontinue drug due to adverse effect | 12 weeks
  Number of participant discontinue drug due to adverse effect wil compared between them

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No